CLINICAL TRIAL: NCT00582751
Title: Volumetric Analysis in the Assessment of Therapy Response by CT
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Robert Lefkowitz, MD, Memorial Sloan-Kettering Cancer Center
Other Study IDs: 07-141; NCT00577291 (obsolete NCT alias)
Record Dates: First submitted 2007-12-21; First posted 2007-12-28 (Estimated); Last update posted 2010-11-02 (Estimated); Status verified 2010-11

CONDITIONS: Multiple Diseases
Keywords: Volumetric Analysis; Multiple Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
To compare the volumetric response achieved using semi-automated computer techniques with the uni-dimensional (RECIST) and bi-dimensional (WHO) criteria as part of clinical trials running at MSKCC, testing new agents for different types of solid tumors.

DETAILED DESCRIPTION:
To compare the volumetric response achieved using semi-automated computer techniques with the uni-dimensional (RECIST) and bi-dimensional (WHO) criteria as part of clinical trials running at MSKCC, testing new agents for different types of solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Registered and being treated on one of the following therapeutic protocols:

06-043, 07-052, 07-057, 07-112, 07-116, 08-093, and 08-054

* Have at least one measurable lesion* as per RECIST criteria situated in lung, liver or lymph node meeting RECIST criteria noted on a baseline CT scan.
* Baseline** and at least one follow-up CT scan to likely to be obtained at an MSKCC facility
* All patients must be > or = to 18 years old

  * The measurable lesions are metastatic in the liver, lung and lymph nodes. The algorithms do not distinguish between primary and metastatic disease, therefore, in selected cases, a primary lesion such as in the liver or lung may also be assessed.

    * Baseline CT are prefer but if not able to obtain for volumetric reconstructions follow up studies will still be use for other objectives if the study.

Exclusion Criteria:

* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 90 patients from 3 different sections will be accrued (30 liver lesions, 30 lung lesions, 30 lymph node lesions).
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2007-11; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
To compare volumetric response achieved using semi-automated computer techniques with the uni-dimensional (RECIST) and bi-dimensional (WHO) criteria as part of clinical trials running at MSKCC, testing new agents for different types of solid tumors. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Robert Lefkowitz, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Web Site — http://www.mskcc.org